CLINICAL TRIAL: NCT04827095
Title: Comparison of Two Web-Based Education/Support Programs for Partner Caregivers of People With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: L-1097-20
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Caregivers; Spouse; Partner; Caregiver Burden; Spinal Cord Injury; Quality of Life; Internet Based Intervention; Grief; Emotions; Clinical Trial
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Support and Education Program 1 (Experimental): The support and education program involves 6 weeks of web-based classes (75-90 minutes per class) given once per week with weekly homework assignments of approximately one hour per week.
  Interventions: Other: Web-Based Support and Education Program 1
- Web-Based Education and Support Program 2 (Experimental): The support and education program involves 6 weeks of web-based classes (75-90 minutes per class) given once per week with weekly homework assignments of approximately one hour per week.
  Interventions: Other: Web-Based Support and Education Program 2

INTERVENTIONS:
Other: Web-Based Support and Education Program 1 — The classes will discuss topics related to caregiving for someone with a spinal cord injury. During these classes, participants will be given information by the class instructor and will also participate in discussions and other learning activities with the rest of the group. Participants will be assigned activities to complete at home for about one hour per week that relate to the topics discussed in class.
  Arms: Web-Based Support and Education Program 1
Other: Web-Based Support and Education Program 2 — The classes will discuss topics related to caregiving for someone with a spinal cord injury. During these classes, participants will be given information by the class instructor and will also participate in discussions and other learning activities with the rest of the group. Participants will be assigned activities to complete at home for about one hour per week that relate to the topics discussed in class.
  Arms: Web-Based Education and Support Program 2

SUMMARY:
The purpose of this research study is to compare the effect of two different types of education and support programs for partner caregivers of people with spinal cord injury (SCI).

DETAILED DESCRIPTION:
SCI particularly affects partners (spouses or other types of significant others), as they face changes in relationship dynamics and identity as they take on a caregiver role. The purpose of this research study is to compare the effect of two different types of education and support programs for partner caregivers of people with spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent in English (reading and writing)
* Romanic partner of a person with SCI (regardless of martial status) for at least one year prior to injury
* Live in a private residence with their partner with SCI
* Partner is at least 3 months post discharge from inpatient rehabilitation
* At least 6 months since their partner's injury
* Provide care to their partner with SCI on a daily basis
* Have access to the internet in a private location

Exclusion Criteria:

* Participant reports a diagnosis of a schizoaffective disorder, bipolar personality disorder, or severe depression
* History of hospitalization for depression treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-29 (Estimated); Study Completion 2023-04-29 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Inhibition/ Behavioral Activation Scale (BIS/BAS) score | Average scores obtained during baseline (pre-program) compared to scores obtained immediately after program completion.
  Change in behavior and emotion, measured by the Behavioral Inhibition/ Behavioral Activation Scale. The extent to which behavior and emotions change over time will be measured with the Behavioral Inhibition/ Behavioral Activation Scale. The BIS/BAS scale is composed of three subscales; (1) drive, which measures the persistent pursuit of goals, (2) fun seeking, which measures the desire for new rewards and the willingness to approach a potentially rewarding event, and (3) reward responsiveness, which measures positive responses to rewarding outcomes.

SECONDARY OUTCOMES:
Change in Marit-Meuser Caregiver Grief Inventory (CGI) scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  50-item inventory scored on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree," used to assess grief before and after participation in the program.
Change in Satisfaction with Life Scale scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  5-item measure of the concept of global life satisfaction before and after participation in the program.
Change in Zarit Burden Interview (ZBI) scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  22-item questionnaire that assesses caregivers' perceptions of burden before and after participation in the program.
Changs in Duke Social Support Index (DSSI) scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  11-item short form that assesses perceived support and non-support from various people in life before and after participation in the program.
Change in Patient Health Questionnaire scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  A self-report questionnaire with subscales for depression and anxiety-related symptoms before and after participation in the program.
Change in NIH Toolbox Loneliness Survey (Fixed Form) scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  Self-report measure of perceptions of loneliness using a 5-item fixed length form before and after participation in the program.
Change in Connor-Davidson Resilience Scale scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  10-item self-report instrument that assesses resilience before and after participation in the program.
Change in Couples Satisfaction Index scores | End of program versus baseline; 3-months post intervention versus baseline, 6-months post intervention versus baseline
  8-item self-report questionnaire assessing perceived strength, comfort, reward, happiness, warmth of relationship to one's partner before and after participation in the program.
Long-Term Change in Behavioral Inhibition/ Behavioral Activation Scale (BIS/BAS) score | 3-months post intervention versus baseline, 6-months post intervention versus baseline
  Change in behavior and emotion, measured by the Behavioral Inhibition/ Behavioral Activation Scale. The extent to which behavior and emotions change over time will be measured with the Behavioral Inhibition/ Behavioral Activation Scale. The BIS/BAS scale is composed of three subscales; (1) drive, which measures the persistent pursuit of goals, (2) fun seeking, which measures the desire for new rewards and the willingness to approach a potentially rewarding event, and (3) reward responsiveness, which measures positive responses to rewarding outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Zanca, PhD, MPT, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No